CLINICAL TRIAL: NCT01050166
Title: Phase 1 Study to Test Safety and Efficacy of Magnetic Resonance Imaging of Human Labeled Islets Transplanted Into the Liver in Type 1 Diabetic Recipients
Brief Title: MRI Imaging of Labeled Human Islets Transplanted Into the Liver
Status: Completed | Type: Observational
Sponsor: Frantisek Saudek (Other Government)
Responsible Party: Sponsor-Investigator, Frantisek Saudek, MD., prof., Institute for Clinical and Experimental Medicine
Organization: Institute for Clinical and Experimental Medicine (Other Government)
Other Study IDs: CD MRI IKEM 1
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: islet transplantation; magnetic resonance; Type 1 DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Labeled islets: Type 1 diabetic recipients after islet transplantation with islets labeled by iron contrast agent
  Interventions: Other: Transplantation of labeled islets

INTERVENTIONS:
Other: Transplantation of labeled islets

SUMMARY:
The purpose of the study is to determine whether human islets labeled by iron contrast agents could be imaged using magnetic resonance after transplantation into the liver of Type 1 diabetic recipients.

DETAILED DESCRIPTION:
Islet transplantation represents approved therapeutic approach in selected Type 1 diabetic recipients with syndrome of hypoglycaemia unawareness. Existing imaging methods are not sufficient to provide adequate information about amount and fate of islets transplanted into the liver. Labeling of islets with superparamagnetic contrast agent ferucarbotran significantly shortens T2 relaxing time and therefore increase the contrast between islets and liver tissue in magnetic resonance imaging. In consequence, islets transplanted into liver could be easily detectable like hypotensive areas dispersed throughout the liver. MRI examination will be done on 1, 2, 4 weeks and 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* normal renal parameters
* hypoglycaemia unawareness or rapid progression of diabetic retinopathy or neuropathy

Exclusion Criteria:

* acute and chronic liver disease
* malignancy
* acute infection
* serious cardiovascular disease
* coagulopathy
* portal hypertension
* presence of metal protesis, cardio-stimulators, or other metal material in the body

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort will be selected from residents of Czech republic
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2008-08-15; Primary Completion 2012-12-15 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Evidence of safety and efficacy of MRI imaging of transplanted human labeled islets | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frantisek Saudek, MD, DrSc, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Diabetes Center, Institute for Clinical and Experimental Medicine, Prague, Czechia

REFERENCES:
- [Result] Saudek F, Jirak D, Girman P, Herynek V, Dezortova M, Kriz J, Peregrin J, Berkova Z, Zacharovova K, Hajek M. Magnetic resonance imaging of pancreatic islets transplanted into the liver in humans. Transplantation. 2010 Dec 27;90(12):1602-6. doi: 10.1097/tp.0b013e3181ffba5e. PMID 21197715